CLINICAL TRIAL: NCT06692075
Title: Emergency Total Extracorporeal Life Support Versus Standard Advanced Cardiac Life Support With ECMO Bailout for Survival With Favorable Neurological Outcome in Refractory Out-of-Hospital Cardiac Arrest
Brief Title: Emergency Total ECLS vs Standard ACLS With ECMO Bailout for Survival in Refractory OHCA
Acronym: ECLS-OHCA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N202312122
Record Dates: First submitted 2024-09-15; First posted 2024-11-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-09

CONDITIONS: Out-of-hospital Cardiac Arrest (OHCA)
Keywords: out-of-hospital cardiac arrest; extracorporeal life support; advanced cardiac life support; sudden death
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Death, Sudden | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Intervention Model Description: Two arms are designed. One is the total ECLS arm to start emergency ECMO supported cardiopulmonary resuscitation immediately after the arrival of eligible OHCA patients at the emergency department. The other is the standard ACLS arm to start standard ACLS cardiopulmonary resuscitation for at least 45 minutes from collapse and 119 call or at least 15 minutes after arrival at the emergency department.
Masking Description: Data and Safety Monitoring Committee
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Total ECLS in refractory OHCA (Active Comparator): Emergency total extracorporeal life support ( ECLS ) in cardiopulmonary resuscitation of OHCA patients with refractory ventricular fibrillation or pulseless ventricular tachycardia
  Interventions: Procedure: extracorporeal life support
- standard ACLS in refractory OHCA (Active Comparator): Emergency standard advanced cardiac life support ( ACLS ) in cardiopulmonary resuscitation of OHCA patients with refractory ventricular fibrillation or pulseless ventricular tachycardia. Bailout ECMO allowed after at least 45 minutes of CPR since collapse and 119 call or at least 15 minutes since arrival at emergency department
  Interventions: Procedure: standard ACLS

INTERVENTIONS:
Procedure: extracorporeal life support — ECMO supported life support for cardiopulmonary resuscitation in refractory OHCA
  Arms: Total ECLS in refractory OHCA
Procedure: standard ACLS — Standard ACLS in cardioplumonary resuscitation of refractory OHCA
  Arms: standard ACLS in refractory OHCA

SUMMARY:
The goal of the clinical trial is to learn if early extracorporeal life support ( ECLS ) will save more out-of-hospital cardiac arrest ( OHCA ) patients with good neurological outcome. It will also learn if emergency ECLS is safe in the OHCA rescue. Researchers aim to investigate if emergency total ECLS is better than standard advanced cardiac life support ( ACLS ) first, followed by bailout ECMO if required, for survival with favorable neurological outcome in OHCA patients. Participants meeting criteria of OHCA with witness, bystander CPR, shockable initial rhythm with repeated defibrillation, and transport time less than 30 min will be compared between total ECLS versus standard ACLS first with bailout ECMO protocols. All participants will receive emergency interventional coronary revascularization , intensive care unit therapy , cardiac ward care and up to 180 days of clinical follow up after survival .

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest ( OHCA ) is a highly lethal emergency, unless return of spontaneous circulation ( ROSC ) is timely achieved by efficient and effective resuscitation. Nevertheless, despite advanced cardiopulmonary resuscitation ( CPR ) with mechanical chest compression, assisted ventilation and automatic external defibrillation, the survival of OHCA patients remains below 10%. Extracorporeal membranous oxygenation ( ECMO ) facilitated life support ( ECLS ) could help hemodynamic stability and improve significantly the survival of refractory OHCA to 25-40 %. On the other hand, the precise role and timing of the ECLS during the emergency management of OHCA remains largely unestablished.

In the present study, we hypothesized that emergency total ECLS is superior to standard ACLS with ECMO bailout for survival with favorable neurological outcome in refractory out-of-hospital cardiac arrest. All OHCA patients meeting the including criteria, i.e. age 18-75 years, witnessed cardiac arrest with bystander CPR, initial shockable rhythm as ventricular fibrillation or pulseless ventricular tachycardia ( VF/pVT ), repeated defibrillation shocks and escorted transportation within 30 minutes from 119 call to arriving emergency department ( ED ) in the hospital would be recruited. Eligible patients will be consecutively randomized at ED in 1:1 ratio, stratified by hospitals, into emergency total ECLS group and standard ACLS with ECMO bailout group. Informed consent is waived in the life-threatening emergency condition. For emergency total ECLS group, OHCA patients will receive early implantation and initiation of ECMO circulation within 15 minutes after randomization or up to 45 minutes after 119 call. For standard ACLS with ECMO bailout group, OHCA patients will receive standard ACLS for at least 45 minutes after collapse or 119 call or at least 15 minutes after ED arrival before calling for bailout ECMO if required. Following return of spontaneous systemic circulation (ROSC) or depending on ECMO circulation, both groups would be transferred to brain and chest computer tomography screening, emergency coronary revascularization intervention and subsequent intensive cardiac care with targeted hypothermia management. Survivals will be treated with guideline directed medical therapy for reduced ejection fraction heart failure and/or implantable cardioverter-defibrillator implantation for prevention of recurrent VT/VF in wards. All survivals will be followed up for medical and neurological status at 30 days, 90 days and 180 days after discharge.

Primary endpoint is survival with favorable neurological outcome at 30 days. Secondary endpoints are survival to discharge with favorable neurological outcome, survival with favorable neurological outcome at 180 days, total duration of cardiopulmonary resuscitation ( CPR ), total duration of mechanical ventilation, total duration of intensive care unit stay, total duration of hospitalization. Safety endpoints will be incidence of serious adverse events related to prolonged CPR, prolonged ischemia, and ECMO systemic perfusion and coronary reperfusion.

The number of subjects to be enrolled according to the primary endpoint of 30 days survival with favorable neurological outcome. With a power of 80%, accepting the level of statistical significance at alpha= 0.05 and based on two-sided Chi-Square test, we estimated 166 participants per arm are needed. This is based on the 30% success rate and 15% success rate of 30-day survival with good neurological outcome of emergency total ECLS intervention and standard ACLS with bailout ECMO (if required) intervention, according to previous trials, plus a 10% drop out rate. Based on two-tailed test, p less than 0.05 is considered statistical significance. If interim analysis is deemed necessary, the significance level will be adjusted accordingly using Bonferroni method. Because of no interim analysis and no stopping point in ITT protocol, there is no criteria for premature termination of the trial. The missing data of the primary and secondary efficacy outcomes will be considered as failure for ITT analysis. Last observations carry forward method will be adapted for the missing data of repeated measurements. The data record will be monitored and audited by the Institutional Review Board of the TMU Shuangho hospital as well as the Data and Safety Monitoring Plan committee.

ELIGIBILITY:
Inclusion Criteria:

1. adults aged 18-75 years old
2. witnessed cardiac arrest with bystander CPR
3. initial shockable rhythm as ventricular fibrillation or pulseless ventricular tachycardia ( VF/pVT )
4. repeated defibrillation shocks ( more than 2 ) by external defibrillator
5. estimated transportation time from 119 call to arrival at emergency service less than 30 minutes.

Exclusion Criteria:

1. age less than 18 years or more than 75 years old
2. non-shockable initial rhythm, i.e. pulseless electrical activity or asystole
3. acute aortic dissection
4. acute massive pulmonary embolism
5. intracerebral hemorrhage
6. major trauma due to blunt, penetrating or burn injury
7. severe peripheral artery occlusion disease
8. known pregnancy
9. suicide, illicit drug overdose or intoxication
10. known pre-arrest modified Rankin score ( mRS ) more than 3 or cerebral performance category scale ( CPC ) more than 2
11. severe concomitant malignancy with expected life expectancy less than 1 year
12. signed and effective do-not-resuscitation ( DNR ) order
13. absolute contraindications to emergency coronary angiography, including known anaphylactic reaction to angiographic contrast media, acute gastrointestinal bleeding or internal bleeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
The rate of survival with favorable neurological outcome ( modified Rankin score less than 3 or cerebral performance category scale 1 or 2 ) at 30 days after discharge from hospital, in percentage | From randomization to 30 days after survival discharge from hospital
  After survival discharge from hospital, clinical followup at out-patient clinic or by visual phone interview is conducted to assess medical health status as well as neurological status of the patients at 30 days after discharge from hospital. Survival with favorable neurological outcome ( i.e. modified Rankin score less than 3 or cerebral performance category scale 1 or 2 ) is to be measured as percentage of all randomized patients fulfilling inclusion criteria and without any exclusion criteria.

SECONDARY OUTCOMES:
Total duration of cardioplumonary resuscitation from on-site CPR by EMS till the stable ROSC or initiation of ECMO life support or the decease of the subject at emergency department up to 30 days after randomization, in minutes | From the start of on-site CPR by EMS till the return of stable ROSC or the initiation of ECMO life support or the decease of the subject at the emergency department up to 30 days after randomization, in minutes
  total duration of standard cardiopulmonary resuscitation ( CPR ) is counted from the start of on-site CPR by emergency medical service ( EMS ) till the stable return of spontaneous circulation ( ROSC ) or initiation of ECMO life support or the decease of the subject at emergency department ( ED ) up to 30 days after randomization. The measure is in minutes.
The rate of survival with favorable neurological outcome ( modified Rankin score less than 3 or CPC scale 1 or 2 ) from the date of randomization to the date of discharge from hospital up to 180 days after randomization, in percentage | From the date of randomization to the date of discharge from hospital up to 180 days after randomization, in percentage.
  At discharge from hospital, patient status is assessed as survival or mortality. The rate of survival with favorable neurological outcome ( modified Rankin score <3 or CPC scale 1 or 2 ) is counted from the date of randomization to the date of discharge from hospital up to 180 days after randomization. The rate of survival is measured as percentage of total randomization number.
The rate of survival with favorable outcomes ( modified Rankin score less than 3 or cerebral performance category scale 1 or 2 ) at 90 days after discharge from hospital, in percentage | From the date of randomization to 90 days after survival discharge from hospital
  After patients survived and discharged from hospital, clinical followup at out-patient clinic or by visual phone interview is conducted to assess medical health as well as neurological status at 90 days after discharge. The rate of survival with favorable neurological outcome ( i.e. modified Rankin score less than 3 or cerebral performance category scale 1 or 2 ) is measured as percentage of all randomized patients fulfilling inclusion criteria and without any exclusion criteria.
The rate of survival with favorable outcomes ( modified Rankin score less than 3 or cerebral performance category scale 1 or 2 ) at 180 days, in percentage | From enrollment to the end of treatment at 180 days
  After patients discharged from hospital, clinical followup at out-patient clinic or by visual phone interview is conducted to assess medical health as well as neurological status at 180 days after discharge. The rate of survival with favorable neurological outcome ( i.e. modified Rankin score less than 3 or cerebral performance category scale 1 or 2 ) is measured as percentage of all enrolled patients fulfilling inclusion criteria and without any exclusion criteria.
total duration of mechanical ventilation from randomization to discharge from hospital or up to 180 days after randomization , in days | From randomization at the emergency department to discharge from hospital or up to 180 days after randomization
  The total duration of assisted mechanical ventilation by volume cycle or pressure cycled artificial ventilators from randomization at the emergency department to discharge from hospital or up to 180 days after randomization, measured in days.
total duration of stay in intensive care ward from randomization to discharge from hospital or up to 180 days after randomization , in days | From the date of randomization to the date of discharge from hospital or up to 180 days after randomization
  The total duration of stay in intensive care ward from randomization to discharge from hospital or up to 180 days after randomization. The intensive care ward is to provide cardiovascular hemodynamic support, assisted mechanical ventilation, targeted temperature therapy ( if needed ) and infection control, whenever needed. The measure is in days.
total duration of hospitalization from the date of randomization to the date of discharge or up to 180 days after randomization , in days | From the date of randomization to the date of discharge from hospital or up to 180 days after randomization, survived or deceased.
  total duration of stay in the hospital from the date randomization at emergency department to the date discharge from hospital or up to 180 days after randomization, survived or deceased. The measure in in days.

CONTACTS AND LOCATIONS:
Locations (1):
- Shuang Ho Hospital, New Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Fu HY, Liu YH, Li SJ, Chang HC, Liu CC, Lee CM, Huang CY, Hsu CW, Ko CI, Wang YC, Chang WT, Wang TJ, Ong JR, Sun JT, Chen JS, Hsu CY, Jang SJ, Chen YL, Lin YH, Chien CY, Kung YC, Wang TL, Yu HC, Hsu CC, Chao CC, Chen CW, Hsu CY, Hsu SC, Chang TI, Yeh JS, Tsai MS, Wei LY, Chou HW, Wang CH, Chang CH, Chen CL, Tu YK, Lin JL, Chen YS. Emergency total extracorporeal life support versus standard advanced cardiac life support with rescue extracorporeal membrane oxygenation for refractory out-of-hospital cardiac arrest: protocol for the ECLS-OHCA randomized trial. Scand J Trauma Resusc Emerg Med. 2026 Feb 3. doi: 10.1186/s13049-026-01557-w. Online ahead of print. PMID 41630056